CLINICAL TRIAL: NCT00574535
Title: Reproductive Hormones And Pre-Clinical CVD In Women
Brief Title: Reproductive Hormones And Pre-Clinical Cardiovascular Disease (CVD) In Women
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Other Study IDs: IRB 4260
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Heart Disease
Keywords: Reproductive Hormones
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Heart disease is not just the number one killer of women, it is also a leading cause of disability. While it is generally believed that heart disease in women is a disease of old age, the stark reality is that heart disease is responsible for more deaths than breast cancer AT ALL AGES. Also, when young women develop heart disease, they are more likely to die or become disabled than their male peers. Identifying women at risk for heart disease is an important step toward reducing the impact of this disease.

Although women can develop heart disease at any age, most women show signs and symptoms of disease about 10 years after men. For years, it has been thought that the reason for this lag is that women's hearts are protected by estrogen, and that when women go through menopause and lose their natural estrogen, they also lose their protection from heart disease. It has been assumed that if estrogen is replaced then protection will continue. These assumptions have not been proven. In fact, three large, randomized trials have shown no benefit from hormone replacement therapy in women known to have heart disease, and in fact have shown that hormone replacement may be harmful.

To better understand the role of hormones and heart disease, the investigators propose to look at markers of heart disease in healthy women and compare this to their natural hormone levels. One of the markers known to be related to heart disease is carotid artery intima-medial thickness (c-IMT) which can be measured by creating an ultrasound picture of an artery in the neck. The investgators will use c-IMT scans and serum blood samples from women in the NIH-sponsored Los Angeles Atherosclerosis Study (LAAS), a large epidemiologic study that followed participants for 8 years. The proposed study will use risk factor information, serum samples and c-IMT scans collected from the female participants (about 269 women) over the 8 years of follow-up. The total sample size is 269 subjects, each of whom donated 3 blood specimens for the LAAS study. This research will examine those specimens (800 in total). It will also measure other markers of heart disease, including inflammation (hsCRP) and diabetes (insulin and glucose). All information has been obtained and there will be no need to collect additional information from participants nor additional blood specimens.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Females
* 40-60 years of age

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Women in LAAS Study
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 1995-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noel Bairey-Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes